CLINICAL TRIAL: NCT00498524
Title: The Sibling Concordance for Implantable Cardioverter-defibrillator Therapies in Ischemic Cardiomyopathy Study
Brief Title: Risk of Life-threatening Heart Rhythm Disturbances in Siblings
Acronym: SIBFIB
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Jonathan P Piccini, Assistant Professor of Medicine, Duke University
Other Study IDs: Pro00001258
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Defibrillators, Implantable; Myocardial Infarction; Tachycardias, Ventricular
Keywords: implantable cardioverter-defibrillator; ischemic cardiomyopathy; ventricular arrhythmias; sibling concordance
MeSH Terms: conditions — Myocardial Infarction; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Sib who has received an ICD
  Interventions: Device: ICD
- 2: Sib who has not received an ICD
  Interventions: Device: ICD

INTERVENTIONS:
Device: ICD — Received an ICD
  Groups: 1
Device: ICD — Have not received an ICD
  Groups: 2

SUMMARY:
The purpose of this study is to determine if heredity influences the risk of life-threatening heart rhythms (ventricular tachycardia and ventricular fibrillation) after heart attack (myocardial infarction).

DETAILED DESCRIPTION:
Greater than 400,000 persons die suddenly each year in the US. The implantable cardioverter-defibrillator (ICD) has revolutionized the primary prevention of sudden cardiac death (SCD) following myocardial infarction (MI), however, risk stratification remains limited and rests solely on the identification of left ventricular dysfunction. The goal of this study is to determine if genetic factors influence the risk of ventricular arrhythmia remotely after myocardial infarction.

In order to determine if ventricular tachycardia or ventricular fibrillation remotely after MI is a heritable trait, we will conduct a family based case-control sibling study of patients who have received an ICD for ischemic cardiomyopathy. As a first step, we will utilize the GENECARD registry, an existing family linkage study of premature cardiovascular disease, to determine the prevalence of sibling concordance for ICD implantation following MI. Probands and siblings in the GENECARD study will be surveyed regarding their ICD history. The sibling recurrence risk ratio for ICD implantation following MI and subsequent ICD therapies will be used to estimate the sample size required to validate heritability, in a larger patient population. In the validation phase of this protocol, we will use a (1) single healthcare system database (Duke Cardiovascular Databank) and a (2) regional population-based registry, in order to determine concordance for ICD therapies. Patients who agree to participate and provide informed consent will be surveyed regarding their personal ICD history and that of their siblings. The prevalence of ICD therapies will be ascertained in the probands, siblings, and the overall cohort. Sibling concordance for ICD implantation and sibling concordance for subsequent appropriate ICD therapies will be used to determine the sibling recurrence risk ratio for appropriate ICD therapies remotely after MI.

ELIGIBILITY:
Inclusion Criteria:

* patients must be alive
* have a history of coronary artery disease / myocardial infarction
* left ventricular ejection fraction ≤ 35%
* received an implantable cardioverter- defibrillator

Exclusion Criteria:

* nonischemic cardiomyopathy
* Pre-identified hereditary arrhythmia syndrome (e.g. long QT syndrome, Brugada syndrome, etc)
* left ventricular ejection fraction >35%
* no implantable cardioverter-defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-MI population with LV dysfunction and an implantable cardioverter-defibrillator.
Sampling Method: Non-Probability Sample
Enrollment: 2047 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
ICD Discharge | Long-term follow up

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Hranitzky, M.D., Principal Investigator — Duke University; Jonathan P Piccini, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Division of Cardiology - Electrophysiology Section, Durham, North Carolina, United States